CLINICAL TRIAL: NCT04706052
Title: Facial Nerve Morbidity After Superficial Parotidectomy in the Absence of Nerve Conductor: an Experience From a Low Resource Country
Brief Title: Facial Nerve Morbidity After Superficial Parotidectomy in the Absence of Nerve Conductor
Status: Completed | Type: Observational
Sponsor: Liaquat University of Medical & Health Sciences (Other)
Responsible Party: Principal Investigator, Fazila Hashmi, Assistant Professor, Liaquat University of Medical & Health Sciences
Other Study IDs: LUMHS/REC/-12
Record Dates: First submitted 2021-01-09; First posted 2021-01-12 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Facial Nerve Injuries; Adenoma, Pleomorphic
Keywords: Superficial Parotidectomy; Facial Nerve Injuries; Adenoma, Pleomorphic
MeSH Terms: conditions — Facial Nerve Injuries; Adenoma, Pleomorphic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Superficial Parotidectomy Patient: All the patients with pleomorphic adenoma irrespective of age and gender who underwent Superficial parotidectomy
  Interventions: Other: Superficial Parotidectomy

INTERVENTIONS:
Other: Superficial Parotidectomy — Classical procedure for pleomorphic adenoma of the parotid gland is superficial parotidectomy around the world. This study only observed the outcome with reference to facial nerve morbidity

SUMMARY:
In this single-centre, cross-sectional case series, the investigators aim to evaluate the incidence of facial nerve injury in patients undergoing superficial parotidectomy in the absence of nerve conductor. Data to be collected retrospectively from a prospectively maintained database of consecutive patients, at the Department of Surgery, Liaquat University of Medical and Health Sciences Jamshoro, Pakistan. The sample size was calculated as 101.

DETAILED DESCRIPTION:
In this single-centre, cross-sectional case series, the investigators aim to evaluate the incidence of facial nerve injury in partcipants undergoing superficial parotidectomy in the absence of nerve conductor. The institutional Research Ethics Committee has approved the study. Data to be collected retrospectively from a prospectively maintained database, at the Department of Surgery, Liaquat University of Medical and Health Sciences Jamshoro, Pakistan. The data period to be over a period of nine years that is from 1st January 2012 till August 2020. The sample size was calculated using the WHO sample size calculator and taking disease prevalence as 7.1 with CI 95%, which turned out to be 101. All the patients with pleomorphic adenoma irrespective of age and gender were included. To control any chance of bias, one of the members of researchers as part of the team who operated upon these patients. The primary outcome was the incidence of temporary or permanent facial nerve injury, while secondary outcomes were wound infection, seroma, hematoma, Frey's syndrome, salivary fistula and disfigured scar. Temporary facial nerve injury was defined as a feature of facial nerve palsy with full recovery to regular activity within six months. Permanent facial nerve injury was defined as any facial nerve dysfunction lasting beyond six months of operation. The data was recorded on a predesigned Performa, and patients' confidentiality was maintained assigning codes to each case known only to researchers. The data was calculated using SPSS version 23. Values of mean and standard deviation were calculated for continuous variables, whereas frequencies were calculated for categorical data.

ELIGIBILITY:
Inclusion Criteria:

* All the patients with pleomorphic adenoma irrespective of age and gender were included

Exclusion Criteria:

* Patients with recurrent disease or unwilling for participation were excluded

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All the suitable and selected patients consented for surgery with an explanation of procedure-related complications. Superficial parotidectomy was a standard surgical procedure for these selected patients with previously untreated pleomorphic adenoma.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
incidence of temporary or permanent facial nerve injury | 12 months
  Temporary facial nerve injury was defined as a feature of facial nerve palsy with full recovery to regular activity within six months. Permanent facial nerve injury was defined as any facial nerve dysfunction lasting beyond six months of operation.

SECONDARY OUTCOMES:
wound infection | 12 months
  Rate of postoperative surgical site infection will be calculated
seroma | 12 months
  Rate of postoperative formation of seroma (non-infected collection) occurring after superficial parotidectomy will be calculated
hematoma | 12 months
  Rate of postoperative incidence of hematoma/ clot formation at the operative site will be calculated
Frey's syndrome | 12 months
  Frey's syndrome is the result of misdirected regeneration of parasympathetic fibres connecting with regenerating sympathetic nerve leading to facial sweating and flushing during times of eating food. Rate of occurrence of Frey's syndrome will be calculated to understand its incidence.
salivary fistula | 12 months
  Salivary fistula is abnormal communication between skin and remaining gland. Its rate of occurrence will be calculated during postoperative period after superficial parotidectomy.
disfigured scar | 12 months
  The number of participants developing cosmetically bad scar will be notified and data calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Fazila Hashmi, FCPS, Principal Investigator — Liaquat University of Medical and Health Sciences Jamshoro Pakistan
Locations (1):
- Fazila Hashmi, Jāmshoro, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Siddiqui AH, Shakil S, Rahim DU, Shaikh IA. Post parotidectomy facial nerve palsy: A retrospective analysis. Pak J Med Sci. 2020 Jan-Feb;36(2):126-130. doi: 10.12669/pjms.36.2.1706. PMID 32063945
- [Background] Bittar RF, Ferraro HP, Ribas MH, Lehn CN. Facial paralysis after superficial parotidectomy: analysis of possible predictors of this complication. Braz J Otorhinolaryngol. 2016 Jul-Aug;82(4):447-51. doi: 10.1016/j.bjorl.2015.08.024. Epub 2015 Dec 19. PMID 26777078
- [Background] Al-Qahtani KH, AlQahtani FM, Muqat MM, AlQahtani MS, Al-Qannass AM, Islam T, Alharbi J, Sebaih H, Alqarni M, Hakami H. A new landmark for the identification of the facial nerve during parotid surgery: A cadaver study. Laryngoscope Investig Otolaryngol. 2020 Jul 28;5(4):689-693. doi: 10.1002/lio2.431. eCollection 2020 Aug. PMID 32864440
- [Background] Saha S, Pal S, Sengupta M, Chowdhury K, Saha VP, Mondal L. Identification of facial nerve during parotidectomy: a combined anatomical & surgical study. Indian J Otolaryngol Head Neck Surg. 2014 Jan;66(1):63-8. doi: 10.1007/s12070-013-0669-z. Epub 2013 Jul 24. PMID 24605304
- [Background] Gaillard C, Perie S, Susini B, St Guily JL. Facial nerve dysfunction after parotidectomy: the role of local factors. Laryngoscope. 2005 Feb;115(2):287-91. doi: 10.1097/01.mlg.0000154735.61775.cd. PMID 15689752